CLINICAL TRIAL: NCT02988830
Title: Impact of Subcutaneous Electric Lumbar Stimulation on Treatment of Refractory Chronic and Disabling Lumbago
Acronym: IMESCUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/39; 2016-A00991-50 (Other: ANSM)
Record Dates: First submitted 2016-11-30; First posted 2016-12-09 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Pain
Keywords: Subcutaneous stimulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chronic lumbar pain (Experimental)
  Interventions: Device: Subcutaneous Electric Lumbar Stimulation

INTERVENTIONS:
Device: Subcutaneous Electric Lumbar Stimulation

SUMMARY:
The aim of the study is to show that subcutaneous electric lumbar stimulation reduces pain in chronic lumbago after 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* Having given their non-opposition
* Affiliated to a national insurance scheme or beneficiary
* Suffering for more than a year from a chronic, invalidating lumbago that is refractory in several lines of treatments

Exclusion Criteria:

* patients with lumbago that can be surgically handled or which justified a medullary stimulation
* having been operated for the rachis for less than 6 months;
* which cannot for cognitive or cultural reasons contribute to the planned evaluations and to the management of the material (remote control);
* for who the investigator can plan that they cannot be followed during one year from the date of the setting-up (non-observance, planned moving, etc.);
* which present psychological, local or general contraindications to the setting-up of a neurostimulation device (Impossibility to stop anticoagulants or aggregation inhibitors, disturb of the hemostasis, cutaneous infection change on the site of setting-up)
* MRI planned within the next year
* pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Average pain per day on visual analogical scale | 12 months

SECONDARY OUTCOMES:
Douleur neuropathique 4 (DN4) score | 12 months
  DN4 is a French neuropathic pain scale
Average pain per day on visual analogical scale | 15 days
OSWESTRY DISABILITY INDEX | 12 months
36-Item Short Form Health Survey score (SF 36) | 12 months
DALLAS self-questionnaire | 12 months
Tampa scale | 12 months
Questionnaire Hospital Anxiety and Depression scale (HAD) | 12 months
Pain Catastrophizing Scale (PCS) | 12 months
Coping strategies questionnaire (CSQ) | 12 months
Fear Avoidance Belief Questionnaire (FABQ) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie Christine DJIAN, MD, Principal Investigator — Hôpital Foch; Bechir Jarraya, MD, PhD, Study Chair — Hôpital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No